CLINICAL TRIAL: NCT06731842
Title: Molecular PET Imaging and Plasma Biomarkers in Alzheimer´s Disease and Other Neurodegenerative Diseases
Acronym: ROADAD
Status: Enrolling by invitation | Phase: Not Applicable | Type: Interventional
Sponsor: Karolinska Institutet (Other)
Responsible Party: Principal Investigator, Agneta Nordberg, MD PhD Professor, Karolinska Institutet
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: 2023-02649
Record Dates: First submitted 2024-12-09; First posted 2024-12-12 (Actual); Last update posted 2024-12-12 (Actual); Status verified 2024-09

CONDITIONS: Alzheimer´s Disease

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- TAU PET and MRI investigation (Other)
  Interventions: Other: 18F-RO948

INTERVENTIONS:
Other: 18F-RO948 — Tau PET imaging using the tau PET tracer 18F-RO948 in famial and sporadic Alzheimer´s disease

SUMMARY:
Multi-modal PET tracer study with the aim of studying the time course of regional deposition of tau in brain of subjects with high risk of being carriers of autosomal dominant Alzheimer´s disease and sporadic early onset and late onset Alzheimer´s disease patient (EOAD, LOAD) in tertiary memory clinic cohort in relation to MRI brain changes, plasma biomarker levels and cognitive performance.

DETAILED DESCRIPTION:
Multi-PET /MRI studies , fluid biomarkers (CSF, plasma) analysis, neuropsychological testing is performed in subjects carriers and non-carriers of different APP, PS autosomal dominant AD mutatation. Both presymptomatic and symptomatic carriers and non-carriers are recruited (age range -30 to +15 years from first clinical symptoms). For comparison also a group of healthy eldersly as well as patients undergoing memory assessment with diagnosis of mild cognitive impairment (amyloid negative /amyloid positive) and diagnosis sporadic Alzheimer´s diases are recruited from Karolinska memory clinic and undergoing similar Multi-PET/MRI studies , fluid biomarker analysis, neuropsycholigal testing. The aim is to describe the evolution and spreading of tau in brain in Alzheimer continuum and compare with other pathological markers with aim of develop new diagnostic markers and therapeutic targets.

ELIGIBILITY:
Inclusion Criteria: a)belonging to families with known familial form of Alzheimer´s disease b) patient undergoing memory assessent at memory clinic with diagnosis mild cognitive impairment (MCI), Alzheimer´s disease c)healthy elderly cognitive normal

-

Exclusion Criteria:

cancer and other serious disease

Ages: 30 Years to 85 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 100 (Estimated)
Dates: Start 2022-05-15 (Actual); Primary Completion 2027-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
PET measurement of regional tau spreading in brain during Alzheimer continuum | 3 years
  Anaysis of regional deposition of tau in brain

CONTACTS AND LOCATIONS:
Overall Officials: Agneta K NORDBERG, MD PhD, Principal Investigator — Karolinska Institutet
Locations (1):
- Karolinska institutet NVS, Stockholm, Sweden

IPD SHARING:
Plan to Share IPD: No
autosomal dominant AD where mutation status is known for participants